CLINICAL TRIAL: NCT00975026
Title: Measuring the Feasibility and the Effects of Chair Massage on Pain and Discomfort in the Cardiac Sonographer - A Pilot Study
Brief Title: Measuring the Feasibility and the Effects of Chair Massage on Pain and Discomfort in the Cardiac Sonographer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deborah Engen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-005517
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Overuse Injury; Repetitive Strain Injury
Keywords: Massage; Chair Massage; Pain; Discomfort; Stretching; Stretching Exercises; Sonographer; Cardiac Sonographer
MeSH Terms: conditions — Cumulative Trauma Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Massages (Active Comparator): Chair massage for 30 minutes once a week.
  Interventions: Procedure: Massages ± Stretches
- Massages + Stretches (Active Comparator): Chair massage for 30 minutes once a week in addition to stretching exercises, to be done twice daily for 20 minutes.
  Interventions: Procedure: Massages ± Stretches
- No Intervention (No Intervention)

INTERVENTIONS:
Procedure: Massages ± Stretches — Chair Massage
  Arms: Massages; Massages + Stretches

SUMMARY:
The purpose of this study is to determine whether the effects of chair massage and/or chair massage with stretching may reduce musculoskeletal pain and discomfort related symptoms associated with the job duties of a cardiac sonographer.

DETAILED DESCRIPTION:
Staff performing echocardiography exams work in a physically demanding environment. The physical and psychosocial demands of the work environment place a significant amount of stress on the physical well being of the employee. The nature of the work involved includes repetitive movements and static holds while applying intense pressure. These compounded by a challenging ergonomic work environment, often leads to physical tension, pain, and fatigue. Staff and patient characteristics, in particular obesity, present greater ergonomic challenges. In this setting, optimal ergonomics can be difficult to achieve. Repetitive actions in an ergonomically challenging environment can have an accumulative effect that can lead to injury.

Massage therapy has been noted to decrease levels of anxiety and fatigue which is essential to maintaining efficient care in a dynamic environment. Repetitive use, typically leads to shortened, tight muscles that fatigue over time. Once the massage therapy has released the connective tissue tension and restored muscle imbalances, exercise focused on core, trunk strength and those muscles which oppose the repetitively used muscles can further assist the therapeutic benefits of massage.

The cardiac sonographer is usually sitting and reaching forward or to the side, and the musculoskeletal imbalances show up primarily superior to the hips. Massage Therapy research for alleviating musculoskeletal symptoms has been with the use of table massage whereas chair massage research has focused on gaining physiological benefits. Chair massage therapy impacts the head, back, neck shoulders, arms and hands so does impact the areas of musculoskeletal imbalance of the cardiac sonographer. In addition, a massage chair is easy to set up, does not need a great deal of space, and can be provided in semi-private area, as the participant remains clothed. Chair massage literature to date has focused more on physiological responses and albeit positive, not as much on musculoskeletal responses.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Sonographer that, per their job descriptions, are performing echocardiography exams during the weeks of the massage therapy pilot study.
* Men and Women age 18-65 able to give informed consent.
* Able to speak and understand English
* 8-hour per day shift schedule, Monday through Friday

Exclusion Criteria:

* Individuals that decline to participate in the study.
* Individuals being treated for an acute musculoskeletal symptom.
* Individuals currently on work restrictions.
* Undergoing treatments for malignancy
* Pregnancy (due to this being chair massage)
* Recent head, neck, shoulder or back surgeries
* Pins or joint fusion of the head or neck
* Current sinus infections, earaches, or vascular migraines
* Students

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Assess the ease and feasibility of providing chair massage therapy in a busy echocardiography exam setting. Compare and contrast the level of pain and discomfort in cardiac sonography staff with three groups over three different time frames. | 10 Weeks

SECONDARY OUTCOMES:
Assess the impact on co-workers as massage therapy is provided during the workday and its effects on workflow. | 10 Weeks
Compare the level of fatigue, stress, anxiety, and relaxation in cardiac sonography staff in each of the 3-arms of the study. | 10 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Engen, O.T., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Engen DJ, Wahner-Roedler DL, Nadolny AM, Persinger CM, Oh JK, Spittell PC, Loehrer LL, Cha SS, Bauer BA. The effect of chair massage on muscular discomfort in cardiac sonographers: a pilot study. BMC Complement Altern Med. 2010 Sep 16;10:50. doi: 10.1186/1472-6882-10-50. PMID 20846441